CLINICAL TRIAL: NCT04735731
Title: Assessing the DIAphragM Before ANd After Endobronchial Valve Treatment
Acronym: DIAMANT
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Dirk-Jan Slebos, MD PhD, University Medical Center Groningen
Other Study IDs: DIAMANT-study
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Emphysema
MeSH Terms: conditions — Emphysema | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EBV-patients: Patients who are scheduled for a bronchoscopic lung volume reduction treatment using endobronchial valves
  Interventions: Diagnostic Test: Echography

INTERVENTIONS:
Diagnostic Test: Echography — Echography of diaphragma and other respiratory muscles

SUMMARY:
Rationale:

The diaphragm is the principal respiratory muscle, which separates the thorax from the abdomen. Hyperinflation of the lung places the diaphragm at a mechanical disadvantage, shortens its operating length and changes the mechanical arrangement of costal and crural components of the diaphragm and consequently decrease the tension that can be developed and the amount of transdiaphragmatic pressure that can be produced. Reducing the lung hyperinflation could improve the diaphragm function mechanically. One of the treatments to reduces lung hyperinflation is the bronchoscopic treatment using endobronchial valves. To our knowledge the change in diaphragm function after bronchoscopic endobronchial valve treatment was never investigated.

Objective:

To investigate the change in diaphragm function after bronchoscopic lung volume reduction treatment with endobronchial valves (EBV).

Study design:

Observational study in which the study population will be asked to perform some additional test during regular visits for the bronchoscopic lung volume reduction treatment with valves.

Main study parameters: Change in diaphragm function 6 week after EBV treatment measured by ultrasound. The main outcome will be diaphragm motion (difference between maximum in- and expiration).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is scheduled for a bronchoscopic lung volume treatment using one-way valves
2. Patient read, understood and signed the Informed Consent Form

Exclusion Criteria:

There are no exclusion criteria for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe emphysema who undergo a bronchoscopic lung volume reduction treatment with one-way endobronchial valves.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2023-01-28 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-02-13 (Actual)

PRIMARY OUTCOMES:
Change in diaphragm motion measured by ultrasound | 6 weeks
  Change in diaphragm motion 6 week after EBV treatment measured by ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk-Jan Slebos, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- UMCG Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Data can be shared on reasonable request